CLINICAL TRIAL: NCT02014103
Title: Evaluation of Clinical and Safety Outcomes Associated With Conversion From Brand-Name to Generic Tacrolimus Products in High Risk Transplant Recipients
Brief Title: Conversion From Brand to Generic Tacrolimus in High Risk Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: University of Colorado, Denver (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Rita Alloway, Research Professor, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13-223-SOL-00102; FDA (Other Grant/Funding Number: HHSF223201310224C)
Record Dates: First submitted 2013-10-21; First posted 2013-12-18 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Complication of Transplant
Keywords: bioequivalence; tacrolimus; transplant; CYP3A5 expressors/non expressors
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Active Comparator): Patients will be randomized to a sequence of administration of the various 6 tacrolimus formulations. Sequence 1: Formulation Sandoz, Panacea, Accord, Mylan, Dr. Reddy's, Astellas
  Patients will be receiving the same tacrolimus dose identified at baseline for each formulation.
  Interventions: Drug: Prograf; Drug: Tacrolimus, Sandoz; Drug: Tacrolimus, Reddy Laboratory; Drug: Tacrolimus, Mylan; Drug: Tacrolimus, Accord; Drug: Tacrolimus, Pancea Biotech Limited
- Sequence 2 (Active Comparator): Patients will be randomized to a sequence of administration of the various 6 tacrolimus formulations. Sequence 2: Formulation Accord, Sandoz, Dr. Reddy's, Panacea, Astellas, Mylan
  Patients will be receiving the same tacrolimus dose identified at baseline for each formulation.
  Interventions: Drug: Prograf; Drug: Tacrolimus, Sandoz; Drug: Tacrolimus, Reddy Laboratory; Drug: Tacrolimus, Mylan; Drug: Tacrolimus, Accord; Drug: Tacrolimus, Pancea Biotech Limited
- Sequence 3 (Active Comparator): Patients will be randomized to a sequence of administration of the various 6 tacrolimus formulations. Sequence 3: Formulation Dr. Reddys, Accord, Astellas, Sandoz, Mylan, Panacea
  Patients will be receiving the same tacrolimus dose identified at baseline for each formulation.
  Interventions: Drug: Prograf; Drug: Tacrolimus, Sandoz; Drug: Tacrolimus, Reddy Laboratory; Drug: Tacrolimus, Mylan; Drug: Tacrolimus, Accord; Drug: Tacrolimus, Pancea Biotech Limited
- Sequence 4 (Active Comparator): Patients will be randomized to a sequence of administration of the various 6 tacrolimus formulations. Sequence 4: Formulation Astellas, Dr. Reddy's, Mylan, Accord, Panacea, Sandoz
  Patients will be receiving the same tacrolimus dose identified at baseline for each formulation.
  Interventions: Drug: Prograf; Drug: Tacrolimus, Sandoz; Drug: Tacrolimus, Reddy Laboratory; Drug: Tacrolimus, Mylan; Drug: Tacrolimus, Accord; Drug: Tacrolimus, Pancea Biotech Limited
- Sequence 5 (Active Comparator): Patients will be randomized to a sequence of administration of the various 6 tacrolimus formulations. Sequence 5: Formulation Mylan, Astellas, Panacea, Dr. Reddy's, Sandoz, Accord
  Patients will be receiving the same tacrolimus dose identified at baseline for each formulation.
  Interventions: Drug: Prograf; Drug: Tacrolimus, Sandoz; Drug: Tacrolimus, Reddy Laboratory; Drug: Tacrolimus, Mylan; Drug: Tacrolimus, Accord; Drug: Tacrolimus, Pancea Biotech Limited
- Sequence 6 (Active Comparator): Patients will be randomized to a sequence of administration of the various 6 tacrolimus formulations. Sequence 6: Formulation Panacea, Mylan, Sandoz, Astellas, Accord, Dr. Reddy's
  Patients will be receiving the same tacrolimus dose identified at baseline for each formulation.
  Interventions: Drug: Prograf; Drug: Tacrolimus, Sandoz; Drug: Tacrolimus, Reddy Laboratory; Drug: Tacrolimus, Mylan; Drug: Tacrolimus, Accord; Drug: Tacrolimus, Pancea Biotech Limited

INTERVENTIONS:
Drug: Prograf — Administration of each formulation will be determined by sequence.
Drug: Tacrolimus, Sandoz — Administration of each formulation will be determined by sequence.
  Other Names: Sandoz tacrolimus
Drug: Tacrolimus, Reddy Laboratory — Administration of each formulation will be determined by sequence.
  Other Names: Reddy's Laboratory tacrolimus
Drug: Tacrolimus, Mylan — Administration of each formulation will be determined by sequence.
  Other Names: Mylan tacrolimus
Drug: Tacrolimus, Accord — Administration of each formulation will be determined by sequence.
  Other Names: Accord Healthcare tacrolimus
Drug: Tacrolimus, Pancea Biotech Limited — Administration of each formulation will be determined by sequence.
  Other Names: Panacea Biotech Limited tacrolimus

SUMMARY:
The prospective study will compare the relative bioavailability at steady-state pharmacokinetics of 6 tacrolimus formulations in a prospective, 6-way cross-over study including CYP3A5 expressors (n=30) and non-expressor (n=30) transplant patients.

DETAILED DESCRIPTION:
Comparison of the relative bioavailability and steady-state pharmacokinetics of 6 tacrolimus formulations in a prospective, 6-way cross-over study including CYP3A5 expressors (n=30) and non-expressor (n=30) transplant patients. Six tacrolimus formulations will be tested and each patient will receive each formulation once. As we proposed to test bioequivalence in the steady-state, patients will receive the test formulations for one week prior to pharmacokinetic evaluation. The pharmacokinetic evaluation will incorporate limited sampling strategies with a focus on fully characterizing the Cmax out to hour 4 post dose. Subsequent PK sampling and trough blood concentrations will be monitored on a daily basis using dried blood spots that the study subjects will collect by themselves at home. It will be critical that the patients are adherent to their test medication to ensure that they have reached steady state. This will be monitored using test diaries, pill counts and MEMS caps (Medication Event Monitoring System (MEMS), AARDEX Corp, Palo Alto, CA. Bioequivalence will be tested using average bioequivalence metrics. A combination of limited sampling strategy and dry spot analysis in combination with population pharmacokinetic modeling will be utilized to fully characterize the PK profile of these formulations.

ELIGIBILITY:
Inclusion criteria

1. 18 years or older
2. Able to participate and willing to give written informed consent/ assent/ consent by parent or legal guardian and to comply with the study visits and restrictions.
3. Subject who has received a primary or secondary transplant.
4. Subject who is at least 6 months post-transplant and on a stable dose of tacrolimus as defined by physician, one tacrolimus trough level within the physician defined target range within past 6 months and one additional trough level during the screening period within 30% of the physician defined target range.
5. BMI less than or equal to 40.

Exclusion criteria

1. Evidence of any acute rejection
2. Subjects who require dialysis within 6 months prior to study entry
3. Recipients of multiple organ transplants
4. Subjects who have tested positive for HBsAG or HIV, or who are recipients of organ from donors who are known to be HBsAG or HIV positive. Virology screening at the time of transplant.
5. HepC positive subjects with liver biopsy proven recurrent disease considered relevant by physician oversight.
6. Subjects with any severe medical condition requiring acute or chronic treatment that in the investigator's opinion would interfere with study participation
7. History of malignancy, treated or untreated, with the past 2 years with the exception of carcinoma in situ or excised basal cell carcinoma, or hepatocellular carcinoma prior to transplant.
8. GFR ≤ 35 ml/min measured as estimated using the MDRD4 formula
9. Subjects with AST, ALT, total bilirubin ≥ 3 X ULN or other evidence of severe liver disease
10. Subjects with white blood cell (WBC) count ≤2,000/ mm3 or with thrombocytopenia (platelet count ≤ 75,000/ mm3), with an absolute neutrophil count of ≤ 1,500/ mm3 or hemoglobin <8g/dL)
11. Subjects with clinically significant infections, requiring therapy, which, in the investigator's opinion, would interfere with the objectives of the study
12. Other mental or physical conditions which in the investigator's opinion, are considered clinically significant
13. Presence of intractable immunosuppressant complications or side effects resulting in dose adjustment of tacrolimus
14. Subjects who have been exposed to an investigational therapy within 30 days prior to enrollment or 5 half-lives of the investigational product, whichever is greater.
15. An anticipated change in the immunosuppressive regimen during subject participation other than that required by the protocol
16. Subject with severe GI disturbance or diarrhea which could interfere with tacrolimus absorption
17. Severe diabetic gastroparesis
18. Initiation of any medications that could interfere with tacrolimus blood levels, including OTC medications, herbal supplements, grapefruit or grapefruit juice.
19. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive BhCG laboratory test (> 5 mIU/mL)
20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are: 1) women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner; 2)women whose partners have been sterilized by vasectomy or 3)using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices (IUDs); periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita R Alloway, PharmD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Expressors: Subjects with at least one *1 allele of CYP3A5
- Non-expressors: Subjects homozygous for the *3 CYP3A5 allele
Period: Overall Study
Arm/Group | Expressors | Non-expressors
Started | 35 | 36
Did Receive Allocated Intervention (One patient did not receive intervention due to elevated SrCr at baseline) | 34 (One patient did not receive intervention due to elevated SrCr at baseline) | 36
Discontinued Intervention | 6 (6 interventions were discontinued. 5 due to protocol defined medication non adherence and one due to lack of venous access) | 5 (5 discontinued intervention Patient unable to complete PK due to personal reasons (2), tacrolimus dose adjustment required during PK (2), and protocol defined nonadherence (1))
Number Subjects Receiving Accord (Subjects were randomized to a sequence of formulation administration for each period. Subjects were withdrawn or dropped out at various periods of the study. The subjects who received identified formulation during the study period of participation are counted.) | 34 | 34
Number Subjects Receiving Astellas (Subjects were randomized to a sequence of formulation administration for each period. Subjects were withdrawn or dropped out at various periods of the study. The subjects who received identified formulation during the study period of participation are counted.) | 32 | 33
Number Subjects Receiving Dr. Reddy (Subjects were randomized to a sequence of formulation administration for each period. Subjects were withdrawn or dropped out at various periods of the study. The subjects who received identified formulation during the study period of participation are counted.) | 34 | 33
Number Subjects Receiving Mylan (Subjects were randomized to a sequence of formulation administration for each period. Subjects were withdrawn or dropped out at various periods of the study. The subjects who received identified formulation during the study period of participation are counted.) | 32 | 34
Number Subjects Receiving Panacea (Subjects were randomized to a sequence of formulation administration for each period. Subjects were withdrawn or dropped out at various periods of the study. The subjects who received identified formulation during the study period of participation are counted.) | 33 | 33
Number Subjects Receiving Sandoz (Subjects were randomized to a sequence of formulation administration for each period. Subjects were withdrawn or dropped out at various periods of the study. The subjects who received identified formulation during the study period of participation are counted.) | 34 | 32
Excluded From Analysis | 2 (Two were excluded from analysis for nonadherence within 48hr of PK visit) | 4 (4 were excluded from analysis. One dure to nonadherence within 48hour of PK visit and 3 due to drug interactions during study period)
Completed | 26 | 27
Not Completed | 9 | 9
Not completed — Protocol Violation | 7 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Lost venous access | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Expressors | Non-expressors | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.5 [46.0 to 62.0] | 57 [44.0 to 62.0] | 56.25 [44 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 1 | 13
  White | 14 | 26 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Compare AUC 0-12hr of Each Tacrolimus Formulation in Expressor and Non Expressor Transplant Recipients
Description: Report the geometric mean and 95% confidence interval for AUC 0-12hr (ng*hr/ml) for each formulation in expressor and non expressor transplant recipients
Time Frame: Whole blood samples were collected immediately prior to dosing, at 1, 1.5, 1.75, 2, 2.5, 3 and 4 hours following dosing. Subjects were then instructed to performed fingersticks using dried blood spot cards at 8 and 12 hours post dose.
Measure: Mean (95% Confidence Interval); unit: ng*hr/ml
Arm/Group | Expressors | Non-expressors
Number analyzed (Participants) | 26 | 27
ng*hr/ml
  Accord | 112.35 [95.83 to 131.72] | 92.37 [81.14 to 105.15]
  Astellas | 97.04 [82.77 to 113.77] | 84.16 [73.93 to 95.81]
  Dr. Reddys | 110.63 [85.83 to 117.98] | 83.96 [73.75 to 95.58]
  Mylan | 96.83 [82.59 to 113.53] | 85.53 [75.13 to 97.37]
  Panacea | 100.58 [85.79 to 117.92] | 89.38 [78.51 to 101.75]
  Sandoz | 98.68 [84.17 to 115.70] | 87.60 [76.95 to 99.73]
Statistical Analysis 1: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Astellas Ratio X 100 = 115.78, 90% CI 2-sided [107.04 to 125.22] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 2: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr. Reddys/Astellas Ratio = 103.7, 90% CI 2-sided [95.91 to 112.12] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 3: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Astellas Ratio X 100 = 99.79, 90% CI 2-sided [92.30 to 107.89] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 4: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 and Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Panacea/Astellas Ratio = 103.65, 90% CI 2-sided [95.83 to 112.11] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 5: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 and parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Sandoz/Astellas Ratio X100 = 101.70, 90% CI 2-sided [94.03 to 110.0] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 6: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Dr Reddys Ratio X 100 = 111.64, 90% CI 2-sided [103.26 to 120.70] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 7: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Mylan Ratio X 100 = 116.02, 90% CI 2-sided [107.27 to 125.49] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 8: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Panacea Ratio X 100 = 111.70, 90% CI 2-sided [103.27 to 120.81] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 9: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Sandoz Ratio X 100 = 113.84, 90% CI 2-sided [105.30 to 123.08] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 10: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Mylan Ratio X 100 = 103.92, 90% CI 2-sided [96.08 to 112.40] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 11: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Panacea Ratio x 100 = 100.05, 90% CI 2-sided [92.50 to 108.21] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 12: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Sandoz Ratio X 100 = 101.97, 90% CI 2-sided [94.28 to 110.29] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 13: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Panacea Ratio X 100 = 96.28, 90% CI 2-sided [89.05 to 104.09] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 14: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Sandoz Ratio X 100 = 98.12, 90% CI 2-sided [90.72 to 106.12] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 15: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Panacea/Sandoz Ratio X 100 = 101.92, 90% CI 2-sided [94.27 to 110.19] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 16: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Astellas Ratio X 100 = 109.75, 90% CI 2-sided [100.42 to 119.25] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 17: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Astellas Ratio X 100 = 99.76, 90% CI 2-sided [91.28 to 109.03] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 18: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Astellas Ratio X 100 = 101.63, 90% CI 2-sided [92.99 to 111.06] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 19: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Panacea/Astellas Ratio X 100 = 106.20, 90% CI 2-sided [97.17 to 116.06] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 20: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Sandoz/Astellas Ratio X 100 = 104.09, 90% CI 2-sided [95.25 to 113.75] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 21: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Dr Reddy Ratio X 100 = 110.02, 90% CI 2-sided [100.66 to 120.24] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 22: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Mylan Ratio X 100 = 108.00, 90% CI 2-sided [98.82 to 118.02] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 23: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Panacea Ratio X 100 = 103.34, 90% CI 2-sided [94.56 to 112.94] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 24: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Sandoz Ratio X 100 = 105.44, 90% CI 2-sided [96.48 to 115.23] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 25: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Mylan Ration X 100 = 98.16, 90% CI 2-sided [89.82 to 107.28] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 26: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr. Reddys/Panacea Ratio X 100 = 93.93, 90% CI 2-sided [85.96 to 102.65] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 27: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Sandoz Ratio X 100 = 95.84, 90% CI 2-sided [87.69 to 104.74] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 28: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Panacea Ratio X 100 = 95.69, 90% CI 2-sided [87.56 to 104.58] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 29: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Sandoz Ratio X 100 = 97.63, 90% CI 2-sided [89.34 to 107.71] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 30: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed AUC 0-12 parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Pancea/Sandoz Ratio X 100 = 102.03, 90% CI 2-sided [93.36 to 111.51] — Bioequivalence is established when 90% confidence interval falls within 80-125

2. Primary Outcome: Compare Cmax of Each Tacrolimus Formulation in Expressor and Non Expressor Transplant Recipients
Description: Report the geometric mean and 95% confidence interval for Cmax (ng/ml) for each formulation in expressor and non expressor transplant recipients
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Expressors | Non-expressors
Number analyzed (Participants) | 26 | 27
ng/ml
  Accord | 21.72 [17.43 to 27.07] | 15.07 [13.02 to 17.44]
  Astellas | 15.31 [12.29 to 19.07] | 13.34 [11.53 to 15.44]
  Dr. Reddys | 15.94 [12.79 to 19.86] | 13.58 [11.73 to 15.71]
  Mylan | 17.76 [14.26 to 22.13] | 15.15 [13.09 to 17.53]
  Panacea | 16.67 [13.38 to 20.78] | 13.23 [11.43 to 15.31]
  Sandoz | 14.40 [11.56 to 17.94] | 12.75 [11.02 to 14.76]
Statistical Analysis 1: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Astellas Ratio X 100 = 141.91, 90% CI 2-sided [125.73 to 160.16] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 2: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Astellas Ratio X 100 = 104.13, 90% CI 2-sided [92.33 to 117.45] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 3: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Astellas Ratio X 100 = 116.02, 90% CI 2-sided [102.87 to 130.87] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 4: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Panacea/Astellas Ratio X 100 = 108.92, 90% CI 2-sided [96.51 to 122.94] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 5: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Sandoz/Astellas Ratio X 100 = 94.06, 90% CI 2-sided [83.33 to 106.16] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 6: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Dr. Reddys Ratio X 100 = 136.27, 90% CI 2-sided [120.82 to 153.70] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 7: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Mylan Ratio X 100 = 122.31, 90% CI 2-sided [108.37 to 138.04] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 8: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Panacea Ratio X 100 = 130.28, 90% CI 2-sided [115.43 to 147.04] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 9: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Sandoz Ratio X 100 = 150.88, 90% CI 2-sided [133.77 to 170.18] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 10: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr. Reddys/Mylan Ratio X 100 = 89.75, 90% CI 2-sided [79.52 to 101.30] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 11: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Panacea Ratio X 100 = 95.60, 90% CI 2-sided [84.71 to 107.90] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 12: Comparison: Expressors; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Sandoz Ratio X 100 = 110.72, 90% CI 2-sided [98.10 to 124.96] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 13: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Panacea Ratio X 100 = 106.52, 90% CI 2-sided [94.44 to 120.15] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 14: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Sandoz Ratio X 100 = 123.36, 90% CI 2-sided [109.30 to 139.23] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 15: Comparison: Expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Panacea/Sandoz Ratio X 100 = 115.81, 90% CI 2-sided [102.68 to 130.62] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 16: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Astellas Ratio X 100 = 112.96, 90% CI 2-sided [100.32 to 127.20] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 17: Comparison: Non-expressors; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Astellas Ratio X 100 = 101.75, 90% CI 2-sided [90.37 to 114.57] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 18: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Astella Ratio X 100 = 113.52, 90% CI 2-sided [100.82 to 127.83] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 19: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Panacea/Astellas Ratio X 100 = 99.16, 90% CI 2-sided [88.06 to 111.64] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 20: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Sandoz/Astellas Ratio X 100 = 95.57, 90% CI 2-sided [84.89 to 107.61] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 21: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Dr Reddy Ratio X 100 = 111.01, 90% CI 2-sided [98.59 to 125.00] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 22: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Mylan Ratio X 100 = 99.51, 90% CI 2-sided [88.38 to 112.04] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 23: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Panacea Ratio X 100 = 113.93, 90% CI 2-sided [101.18 to 128.28] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 24: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Accord/Sandoz Ratio X 100 = 118.19, 90% CI 2-sided [104.96 to 133.08] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 25: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr Reddys/Mylan = 89.64, 90% CI 2-sided [79.61 to 100.93] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 26: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr. Reddys/Panacea Ratio X 100 = 102.63, 90% CI 2-sided [91.15 to 115.55] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 27: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Dr. Reddys/Sandoz Ratio X 100 = 106.46, 90% CI 2-sided [94.55 to 119.88] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 28: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Panacea Ratio X 100 = 114.49, 90% CI 2-sided [110.68 to 128.92] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 29: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Mylan/Sandoz Ratio X 100 = 118.77, 90% CI 2-sided [105.48 to 133.74] — Bioequivalence is established when 90% confidence interval falls within 80-125
Statistical Analysis 30: Comparison: Non-expressors; Analysis of variance (PROC MIXED) was performed on log transformed Cmax parameters; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% confidence interval falls within 80-125; Geometric Panacea/Sandoz Ratio X 100 = 103.74, 90% CI 2-sided [92.13 to 116.81] — Bioequivalence is established when 90% confidence interval falls within 80-125

3. Secondary Outcome: To Compare the Safety and Efficacy of Each Tacrolimus Formulation in Stable Transplant Subjects
Description: Conduct safety lab testing specific to transplanted organ function and clinical assessments for adverse events.
Time Frame: Assessed at baseline and weekly for 6 weeks at each pharmacokinetic profile
Population: Participants in the PK population with available data
Measure: Count of Participants; unit: Participants
Groups:
- Accord: Subjects receiving the Accord formulation
- Astellas: Subjects receiving the Astellas formulation
- Dr. Reddys: Subjects receiving the Dr Reddy formulation
- Mylan: Subjects receiving the Mylan formulation
- Panacea: Subjects receiving the Panacea formulation
- Sandoz: Subjects receiving the Sandoz formulation
Arm/Group | Accord | Astellas | Dr. Reddys | Mylan | Panacea | Sandoz
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53 | 53
Participants
  All cause mortality | 0 | 0 | 0 | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Total Other Adverse Events (not including Serious) | 22 | 14 | 20 | 22 | 23 | 13
  Nervous system | 2 | 0 | 2 | 4 | 4 | 1
  Blood and Lymphatic system | 0 | 0 | 1 | 0 | 0 | 0
  Cardiac | 1 | 0 | 1 | 1 | 2 | 1
  Ear and labyrinth | 0 | 1 | 0 | 0 | 0 | 0
  Metabolism and Nutrition | 2 | 1 | 1 | 2 | 4 | 2
  Gastrointestinal | 4 | 1 | 2 | 2 | 2 | 2
  Respiratory, thoracic, and mediastinal | 0 | 1 | 0 | 2 | 1 | 0
  Musculoskeletal and connective tissue | 1 | 1 | 1 | 0 | 2 | 1
  Reproductive system and breast disorders | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations | 0 | 0 | 0 | 1 | 1 | 0
  Skin and subcutaneous tissue | 0 | 1 | 0 | 1 | 0 | 0
  Psychiatric | 0 | 1 | 0 | 0 | 0 | 1
  Vascular | 0 | 1 | 2 | 1 | 1 | 0
  Investigations | 4 | 1 | 1 | 0 | 2 | 1
  Renal and urinary | 1 | 1 | 5 | 1 | 1 | 1
  Allergies | 0 | 1 | 0 | 0 | 0 | 0
  Eye Disorder | 2 | 0 | 1 | 0 | 0 | 1
  Endocrine | 1 | 0 | 0 | 0 | 0 | 0
  General disorders and administrative site conditions | 4 | 3 | 3 | 7 | 3 | 2

ADVERSE EVENTS:
Time Frame: Data was collected during the 6 week period enrolled in the pharmacokinetic study
Arm/Group | Accord | Astellas | Dr. Reddys | Mylan | Panacea | Sandoz
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/53 | 0/53 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/53 | 0/53 | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 22/53 | 14/53 | 20/53 | 22/53 | 23/53 | 13/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accord (N=53) | Astellas (N=53) | Dr. Reddys (N=53) | Mylan (N=53) | Panacea (N=53) | Sandoz (N=53)
Anxiety, tremor (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (7) | 4 (4) | 1 (1)
leukopenia, thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypertension, tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
ear erythemia (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dehydration, hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
nausea, vomitting, diarhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
respiratory tract infections (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
lost venous access (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
study related issues (Investigations) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
difficult urinating (Renal and urinary disorders) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 1 (1)
allergies (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
eye redness, itching (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
administrative issues (General disorders) | 4 (7) | 3 (3) | 3 (4) | 7 (7) | 3 (3) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No